CLINICAL TRIAL: NCT02832440
Title: Comparison of Intradialytic Versus Home-based Programmes on Adherence and Strength of Stage 5 Chronic Kidney Disease Patients
Brief Title: Comparison of Two Exercise Programmes in Patients Undergoing Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU Card Herrera
Record Dates: First submitted 2016-07-08; First posted 2016-07-14 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Intradialytic exercise (Other): Exercise during hemodialysis
  Interventions: Other: Exercise programmes
- Home-based exercise (Other): Exercise at home
  Interventions: Other: Exercise programmes

INTERVENTIONS:
Other: Exercise programmes

SUMMARY:
Although exercise training of haemodialysis patients is associated with generally positive outcomes few haemodialysis units routinely offer intradialytic exercise therapy. This is often related to financial cost and/or staffing limitations. Home-based programs could be an alternative means of providing exercise benefits without associated implementation costs The aim of this study was to compare the effects of 4 weeks intradialytic versus home based exercise for haemodialysis patients regarding adherence and strength gains.

ELIGIBILITY:
Inclusion Criteria:

* people under hemodialysis treatment at least 3 months
* be medicable stable
* complete all the physical tests

Exclusion Criteria:

* heart stroke in the previous 6 weeks of the study
* inferior limb amputation without artificial aids
* cerebral vascular disease (ictus, ischemic)
* disability to complete functional tests

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Short Physical Performance Battery at 4 months | At the beginning and after 4 months
  Assess lower extremity, which includes objective performance-based measure of balance (side-by-side, semi-tandem and tandem), endurance (4m gait speed) and strength (five chair stands). Each component was scored from 0 to 4 and when summed yielded Short Physical Performance Battery scores between 0 (poor) and 12 (best).
Change from Baseline One leg standing test at 4 months | At the beginning and after 4 months
  Consist in maintain one leg stance for as long as possible. The test was considered normal if the one leg standing time reached 45 seconds.
Change from Baseline Timed Up and Go test at 4 months | At the beginning and after 4 months
  To stand up from a standard arms chair, walk 3 meters, turn back the cone walk back and sit down to the chair. The time in seconds is record.
Change from Baseline Sit to stand to sit 10 and 60 at 4 months | At the beginning and after 4 months
  For the Sit To Stand 10 participant has to stand up and sit down 10 times and the time needed is record; while for the Sit to stand to sit 60 the participant consist in measures how many repetition the participant can to stand up and sit down during 60 seconds
Change from Baseline One leg heel rise at 4 months | At the beginning and after 4 months
  It measures the strength in the triceps surae in the one leg standing position and has to rise the heel. It measures how many repetitions the participants is can do
Change from Baseline Handgrip Strength at 4 months | At the beginning and after 4 months
  To measure the amount of strength developed by each hand in kg
Change from Baseline Six minutes walking test at 4 months | At the beginning and after 4 months
  To walk the longest distance possible in 6 minutes by walking continuously the 20 or 30 metres indicated on the floor. It measures the distance in meters

CONTACTS AND LOCATIONS:
Overall Officials: Eva Segura Ortí, Principal Investigator — Lecturer in the Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain